CLINICAL TRIAL: NCT07115745
Title: A Phase 1, Multicenter, Open-label Study of BMS-986515, Healthy Donor Allogeneic CD19-targeted Chimeric Antigen Receptor (CAR) T Cells, in Participants With Severe, Refractory Autoimmune Diseases
Brief Title: A Study of Healthy Donor CD19-targeted Allogeneic CAR T Cells in Participants With Severe, Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM060-0001; 2024-517681-41 (Other: EU CTR); U1111-1308-9273 (Other: WHO)
Record Dates: First submitted 2025-02-07; First posted 2025-08-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Refractory Autoimmune Diseases
Keywords: CAR-T; Cell Therapy; Autoimmune disease; Systemic lupus erythematosus; idiopathic inflammatory myopathy; systemic sclerosis; rheumatoid arthritis; Musculoskeletal Diseases; Myositis; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Scleroderma, Diffuse; Autoimmune Diseases; Sclerosis; Skin Diseases; Connective tissue diseases; BMS-986515; Allogeneic CAR T; CD19 Allogeneic CAR T; AlloCAR T, Cell Therapy; CAR T; SLE; Lupus Nephritis; SSc; IIM; Polymyositis; Dermatomyositis; RA
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Arthritis, Rheumatoid; Musculoskeletal Diseases; Scleroderma, Diffuse; Sclerosis; Skin Diseases; Connective Tissue Diseases; Lupus Nephritis; Polymyositis; Dermatomyositis | interventions — fludarabine; Cyclophosphamide; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986515 Administration (Experimental)
  Interventions: Genetic: BMS-986515; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tocilizumab

INTERVENTIONS:
Genetic: BMS-986515 — Specified dose on specified days
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days
Drug: Tocilizumab — Specified dose on specified days

SUMMARY:
The purpose of this study is to determine the safety, tolerability, optimal dose, and preliminary efficacy of BMS-986515, a healthy donor (HD) allogeneic CD19-targeted CART cell product, in participants with severe, refractory autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria

- Systemic lupus erythematosus (SLE) population:.

i) Diagnosis of SLE based on the 2019 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR).

ii) Participant must be positive for at least one of the following antibodies at screening: anti-nuclear antibody, anti-dsDNA, anti-histone, anti-chromatin or anti-Sm antibody.

iii) Inadequate response or intolerance to steroids and immunosuppressive therapies.

iv) Participants must have active disease at screening.

- Inflammatory myopathy (IIM) population:.

i) Participants meeting the 2017 American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) classification criteria.

ii) Participants must meet criteria for with severe, refractory IIM. iii) Participants who had inadequate response to steroids and prior immunosuppressive therapies.

iv) Evidence of active disease.

- Systemic sclerosis (SSc) population:.

i) Participant must fulfill the 2013 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) classification criteria for systemic sclerosis.

ii) Inadequate disease response or intolerance to prior therapies. iii) Participants diagnosed with progressive systemic sclerosis including skin disease and/or interstitial lung disease.

- Rheumatoid arthritis (RA) population:.

i) Participants with difficult to treat RA. ii) Participants with a diagnosis of RA meeting 2010 ACR/EULAR criteria. iii) Rheumatoid arthritis disease activity at screening and baseline visit. iv) Inadequate disease response or intolerance to standard of care therapy.

Exclusion Criteria

- All participants:.

i) Any other systemic autoimmune disease. ii) Pregnant or nursing women. iii) Active hepatitis B, C or HIV. iv) Prior history of malignancies. v) Uncontrolled or active infection. vi) History of certain cardiovascular conditions within 6 months prior to screening.

vii) Previous CAR-T cell therapy. viii) Significant lung impairment. ix) Inadequate organ function. x) Active, clinically significant, central nervous system (CNS) disorders.

* SLE population:.

  i) Participants who have SLE because of drugs or have other autoimmune diseases along with SLE.
* IIM population:.

  i) Participants who have other forms of myopathies other than IIM. ii) Severe muscle damage.
* SSc population:.

  i) People who have high blood pressure in the arteries of the lungs caused by SSc, which needs regular treatment to keep it under control.

ii) Rapidly deteriorating SSc, or history of severe kidney disease.

* RA population:.

  i) People who have additional autoimmune diseases along with RA.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2029-02-13 (Estimated); Study Completion 2030-08-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 24 months post BMS-986515 infusion
  All participants
Number of participants with serious AEs (SAEs) | Up to 24 months post BMS-986515 infusion
  All participants
Number of participants with AEs of special interest (AESIs) | Up to 24 months post BMS-986515 infusion
  All participants
Number of participants with laboratory abnormalities | Up to 24 months post BMS-986515 infusion
  All participants
Number of participants with Dose-Limiting Toxicities (DLTs) | Up to 24 months post BMS-986515 infusion
  All participants
Number of participants with DLTs that occur during the DLT evaluation period | 28 days post-BMS-986515 infusion
  All participants

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 2 years
  All participants
Area under the concentration-time curve (AUC) | Up to 2 years
  All participants
Time of maximum observed concentration (Tmax) | Up to 2 years
  All participants
Number of participants with interstitial lung disease (ILD) with no worsening of pulmonary function from baseline to Week 24 | Up to 2 years
  All participants
Number of participants who achieve definition of remission in systemic lupus erythematosus (DORIS) remission at Week 24 | Up to Week 24
  Systemic lupus erythematosus (SLE) participants
Number of participants who achieve Lupus Low Disease Activity State (LLDAS) at Week 24 | Up to Week 24
  SLE participants
Change in proteinuria measured by urine protein creatinine ratio (UPCR) from baseline to Week 24 | Up to Week 24
  SLE participants
Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) from baseline to Week 24 | Up to Week 24
  SLE, systemic sclerosis (SSc), and rheumatoid arthritis (RA) participants
Number of participants who achieve Myositis Response Criteria Total Improvement Score (MRC TIS) at Week 24 | Up to Week 24
  Inflammatory myopathy (IIM) participants
Change in International Myositis Outcome Assessment Collaborative Study Group (IMACS) outcome measure set for disease activity at week 24 from baseline | Up to Week 24
  IIM participants
Change in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) at week 24 from baseline | Up to Week 24
  Dermatomyositis (DM) participants only
Number of participants who achieve an minimal clinically important differences in SSc (MCID) from baseline of the modified Rodnan Skin Score (mRSS) at Week 24 | Up to Week 24
  SSc participants
Change from baseline of the Revised Composite Response Index in Systemic Sclerosis (CRISS) at Week 24 | Up to Week 24
  SSc participants
Number of participants with low disease activity at Week 24 from baseline | Up to Week 24
  RA participants

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- United States (3):
  - Local Institution - 0041, Boston, Massachusetts
  - Local Institution - 0037, Durham, North Carolina
  - Local Institution - 0033, Seattle, Washington
- Australia (3):
  - Local Institution - 0007, Camperdown, New South Wales
  - Local Institution - 0008, Brisbane, Queensland
  - Local Institution - 0013, Clayton, Victoria
- Brazil (3):
  - Local Institution - 0040, Salvador, Estado de Bahia
  - Local Institution - 0039, Porto Alegre
  - Local Institution - 0038, São Paulo
- Czechia (2):
  - Local Institution - 0004, Prague, Praha 5
  - Revmatologicky ustav, Prague
- France (2):
  - CHU Strasbourg-Hautepierre, Strasbourg, Alsace
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
- Germany (5):
  - Local Institution - 0023, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Charité - Universitaetsmedizin Berlin - Campus Bejnamin Franklin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Local Institution - 0031, Hamburg
- Israel (2):
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Szpital Specjalistyczny nr 1 w Bytomiu, Bytom, Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy w Gliwicach, Gliwice, Silesian Voivodeship
  - Local Institution - 0017, Lodz, Łódź Voivodeship
- Romania (2):
  - ARENSIA Exploratory Medicine, Cluj-Napoca, Cluj
  - Fundeni Clinical Institute, Bucharest
- Spain (3):
  - Local Institution - 0011, Barcelona, Barcelona [Barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07115745.html